CLINICAL TRIAL: NCT06521333
Title: Efficacy of Resveratrol-Based Gel Versus Hyaluronic Acid Gel as a Palatal Wound Dressing Materials on Postoperative Pain Following Free Gingival Graft Surgery: A Randomized Controlled Clinical Trial
Brief Title: Resveratrol-Based Gel Application in a Palatal Wound Following Free Gingival Graft Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Liza saleh kasem ALhakam, Dentist, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 19424
Record Dates: First submitted 2024-07-21; First posted 2024-07-25 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: Mucogingival Defects
MeSH Terms: interventions — Stents

STUDY DESIGN:
Intervention Model Description: A Randomized Controlled Clinical Trial
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Resveratrol-Based gel (Experimental): The Resveratrol-Based gel will be applied using a sterile plastic syringe, and the palatal wound will be immediately covered by an acrylic resin stent. Three days postoperatively, the patients will be recalled, the stent will be removed for evaluation and the Resveratrol gel will be reapplied.
  Interventions: Drug: Resveratrol-Based gel
- Hyaluronic acid gel 0.2% (Active Comparator): 0.2% hyaluronic acid gel (Gengigel®) The 0.2% Hyaluronic acid gel will be applied using a sterile plastic syringe, and the palatal wound will be covered by an acrylic resin stent. Three days postoperatively, the patients will be recalled, the stent will be removed for evaluation, and the Hyaluronic acid gel will be reapplied.
  Interventions: Drug: Hyaluronic acid gel 0.2%
- Acrylic resin stent only. (Placebo Comparator): The palatal donor site covered with acrylic resin stent only.
  Interventions: Device: Stent

INTERVENTIONS:
Drug: Resveratrol-Based gel — The Resveratrol-Based gel will be applied using a sterile plastic syringe, and the palatal wound will be immediately covered by an acrylic resin stent. Three days postoperatively, the patients will be recalled, the stent will be removed for evaluation and the Resveratrol gel will be reapplied.
  Arms: Resveratrol-Based gel
Drug: Hyaluronic acid gel 0.2% — The 0.2% Hyaluronic acid gel will be applied using a sterile plastic syringe, and the palatal wound will be covered by an acrylic resin stent. Three days postoperatively, the patients will be recalled, the stent will be removed for evaluation, and the Hyaluronic acid gel will be reapplied.
  Other Names: Gengigel
  Arms: Hyaluronic acid gel 0.2%
Device: Stent — The palatal wound will be immediately covered by acrylic resin stent three days postoperatively, the patients will be recalled, and the stent will be removed for evaluating the healing of the palatal wound and then recover with stent.
  Arms: Acrylic resin stent only.

SUMMARY:
Aim of the study to compare the effect of Resveratrol- Based gel versus 0.2% Hyaluronic acid gel applied to the palatal donor site and acrylic resin stent only in post-operative pain reduction after free gingival graft harvesting.

DETAILED DESCRIPTION:
Treatment Protocol Presurgical Phase Initial phase will involve comprehensive periodontal treatment, including full mouth supragingival scaling, subgingival debridement using ultrasonic devices and Gracey curettes, and polishing one month prior to surgery. Patients will receive detailed instructions on mechanical plaque control techniques, such as the brushing technique with a soft toothbrush, and the importance of maintaining oral health.

Additionally, 0.12% Chlorhexidine HCL mouthwash will be prescribed for chemical plaque control, to be used twice daily for 2 weeks.

Surgical procedure Step 1: Preparing the recipient site. Step 2: Harvesting the free gingival graft from palate. The Free Gingival Graft (FGG) will be harvested from the palate using a standardized technique. The palatal sites will be anaesthetized with a solution of 2% lidocaine and 0.001% adrenaline. A partial thickness graft, consisting of epithelium and a thin layer of connective tissue, will be harvested with proper thickness between 1.0 and 1.5 mm for optimal graft survival.

Step 3: Placement of free gingival graft on the recipient beds Step 4: Management of the Palatal Wound

Denuded palatal area will be protected using one of the following options:

1. Resveratrol- Based gel covered with acrylic resin stent (test group I).
2. Hyaluronic acid (HA) gel 0.2% with acrylic resin stent (test group II)
3. Acrylic resin stent (control group III) Test Group I Resveratrol- Based gel The Resveratrol-Based gel will be applied using a sterile plastic syringe, and the palatal wound will be immediately covered by an acrylic resin stent. Three days postoperatively, the patients will be recalled, the stent will be removed for evaluation and the Resveratrol gel will be reapplied. Test Group II (0.2% HA) 0.2% hyaluronic acid gel (Gengigel®) The 0.2% Hyaluronic acid gel will be applied using a sterile plastic syringe, and the palatal wound will be covered by an acrylic resin stent. Three days postoperatively, the patients will be recalled, the stent will be removed for evaluation, and the Hyaluronic acid gel will be reapplied.

Group III (Control Group) The palatal wound will be immediately covered by acrylic resin stent three days postoperatively, the patients will be recalled, and the stent will be removed for evaluating the healing of the palatal wound and then recover with stent.

Step 5: Postoperative care The postoperative instructions will be specified to avoid using a toothbrush or floss in the vicinity of the surgical sites. During the first week, patients will be instructed to limit their food intake to soft foods and to avoid any mechanical trauma.

Patient evaluation of post-operative morbidity and aesthetics will be conducted during appointments on days 3, 7, 14, 21, and 42 following the evaluation.

ELIGIBILITY:
Inclusion Criteria:

1. Patient over 18 years of age
2. Systemically healthy
3. Plaque index (PI) and gingival index (GI) less than 15% (Silness & Löe)
4. Patients with Mucogingival defects scheduled for free gingival graft

Exclusion Criteria:

1. Pregnancy or breastfeeding.
2. Occlusal trauma at site of graft.
3. Severe gagging reflex
4. Smokers.
5. Patients allergic to the used materials.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-05-14 (Actual); Primary Completion 2025-08-30 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative Pain | at (0--7 days)
  direct measure by using Visual Analog Scale (VAS) pain scores (ranging from 0 to 10, where 0 indicates no pain 1: minimal pain and 10 signifies severe pain) will be recorded daily for one week as the pain is expected to reach its maximum level during the initial healing phase (0-3 days)

SECONDARY OUTCOMES:
Indirect Postoperative Pain by analgesic consumption consumption Postoperative | at (0-7) days
  Pain Indirect measurement by analgesic consumption Postoperative for 7 days postoperatively
Wound size | at surgery day, day 3, day 7, day 14 and day 21
  measure by using UNC-15 periodontal probe.
patient satisfaction with the healing process | completed 1 week after the surgery
  measure by using Visual analogue scale.
  a Visual Analog Scale (VAS) specifically designed for measuring patient satisfaction with medical care. This type of scale allows patients to express their level of satisfaction by marking a point along a continuous line, which is typically 10 cm long, representing a range from complete dissatisfaction (0) to full satisfaction (10).
Color match.. | on day 3, day 7, day 14, day 21, and day 42
  measure by using Visual analogue scale. Colour match (CM) of the donor site was also assessment by using VAS scores (between 0 and 10. 0: no CM, 10: excellent CM) in comparison with adjacent and contra-lateral palatal mucosa.

CONTACTS AND LOCATIONS:
Overall Officials: Liza S ALhakam, Principal Investigator — master student.; Manar T El-Zanaty, PhD, Study Chair — Lecturer of oral medicine and Periodontology, Faculty of Dentistry, Cairo University.; Enji A Mahmoud, Professor, Study Director — Professor of Oral Medicine and Periodontology, Faculty of Dentistry, Cairo University.
Locations (1):
- Faculty of dentistry, Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided